CLINICAL TRIAL: NCT04523740
Title: Paracetamol Discontinuation in the Elderly After Long-term Consumption
Acronym: PARADISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Lykke Ida Kaas Oldenburg, MSc Pharm, PhD candidate, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2019-000203-33
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Pain, Chronic; Pain, Medication; Pain, Discontinuation
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo replacement (Experimental): Participants will discontinue the paracetamol treatment, and be administered 6 to 8 tablets of placebo per day
  Interventions: Drug: Placebo
- Usual care with paracetamol (Active Comparator): Participants will continue the paracetamol treatment, and be administered 6 to 8 tablets of 500mg paracetamol per day
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Placebo — Patients who use regular paracetamol will now receive 6 to 8 tablets of placebo per day for 2 weeks
  Arms: Placebo replacement
Drug: Paracetamol — Patients who use regular paracetamol will now receive 6 to 8 tablets of 500 mg paracetamol per day for 2 weeks
  Other Names: Acetaminophen
  Arms: Usual care with paracetamol

SUMMARY:
To investigate if long-term treatment of paracetamol can be discontinued without no worsening on pain, health-related quality-of-life and level of function compared to continuing paracetamol treatment in patients aged 65 years or more.

DETAILED DESCRIPTION:
Aim: To investigate if long-term treatment of paracetamol can be discontinued without worsening on pain, health-related quality-of-life and level of function compared to continuing paracetamol treatment in patients aged 65 years or more.

Trial design: Patients are randomized to either arm 1: standard care (paracetamol continuation) or arm 2: experimental treatment (placebo).

The investigation is double-blinded.

Patients are screened and recruited from Department of respiratory medicine at Copenhagen University Hospital Bispebjerg. Patients with a daily consumption of 3 grams or more of prescribed paracetamol and who comply with the other eligibility criteria will be invited to participate in the trial and asked for written, informed consent. If given we collect data regarding the patient's medications, any medication changes during the intervention and followup, frailty (FRAIL Scale), self-reported history of falls, recent admissions, self-reported health-related quality of life (EQ-5D-5L), level of function tested by hand grib strength and sitting-rising test, and death.

Data is collected at baseline and after 2 weeks when ending treatment intervention, and a 26 week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or more
* Regular daily users of 3 to 4 grams of paracetamol for at least 6 months prior to enrollment

Exclusion Criteria:

* Malignant pain cf. their medical records
* Patients using other regular analgesics cf. indication on prescription
* Patients receiving paracetamol tablets with modified release or sustained release
* Patients in warfarin treatment
* Patients with terminal illnesses, cf. their medical records.
* Patients receiving dosages dispensed by their pharmacy
* Mini-Mental State Examination (MMSE) score less than 25
* Patients with or suspected to have COVID-19.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) pain during til last 24 hours | Change from baseline value at week 2
  Comparison of changes in visual analog scale (VAS) pain intensity during the last 24 hours, from baseline value at week 2 between the control and intervention group. VAS is a 0-100 mm scale where 0 is "no pain" and 100 is "worst pain"

SECONDARY OUTCOMES:
EQ5D-5L index | Change from baseline value at week 2
  Comparison of changes in EQ5D-5L index from baseline values at week 2 between the control and intervention group. EQ-5D is an abbreviation for "European Quality of life - 5 Dimensions" and measures Quality of Life. The scale has five subcomponents with scores from 1 (best) to 5 (worst). The five subcomponents constitute a health state that is translated into an index value using the Danish Crosswalk Index Value Calculator from Euroqol's website. The index value is anchored at 0 = death and 1 = full health and the range in the Danish population is from -0.624 (worse than death) to 1.0 (full health). Higher values / increases in index value is better than lower values / decreases in index value.
Treatment failure. | Week 2
  Number of participants that initiate other regular analgesics or withdraw from the trial
Grip strength | Change from baseline value at week 2
  Functional level is measured by grib strength with a Hand Dynamometer
Sitting-rising test | Change from baseline value at week 2
  Functional level is measured by a sitting-rising test
Sum of daily visual analog scale (VAS) pain | Sum from baseline to week 2
  Collected from a trial diary. Visual analog scale (VAS) is a 0-100 mm scale where 0 is "no pain" and 100 is "worst pain"
Followup: Number of regular users (3 grams of paracetamol or more per day) since ending treatment period. | week 26
  Did the intervention change the participants' paracetamol consumption after ending the treatment period.
Followup: Visual analog scale (VAS) pain during til last 24 hours | Week 26
  Comparison of changes from baseline and week 2 values at week 26 (post treatment period). Visual analog scale (VAS) is a 0-100 mm scale where 0 is "no pain" and 100 is "worst pain"
Followup: EQ5D-5L index | Week 26
  Comparison of changes in EQ5D-5L index from baseline and week 2 values at week 26 (post treatment period) between the control and intervention group. EQ-5D is an abbreviation for "European Quality of life - 5 Dimensions" and measures Quality of Life. The scale has five subcomponents with scores from 1 (best) to 5 (worst). The five subcomponents constitute a health state that is translated into an index value using the Danish Crosswalk Index Value Calculator from Euroqol's website. The index value is anchored at 0 = death and 1 = full health and the range in the Danish population is from -0.624 (worse than death) to 1.0 (full health). Higher values / increases in index value is better than lower values / decreases in index value.
Trial failure | Week 26
  Number of participants who initiated regular use of other analgesics and comparison of changes between the control and intervention group (post treatment period)

CONTACTS AND LOCATIONS:
Overall Officials: Jon T Andersen, MD, PhD, Principal Investigator — Department of Clinical Pharmacology
Locations (1):
- Department of clinical pharmacology, Copenhagen, Bispebjerg, Denmark

IPD SHARING:
Plan to Share IPD: No